CLINICAL TRIAL: NCT01130181
Title: Correction of Vitamin D Deficiency in Critically Ill Patients: a Randomized, Double-blind, Placebo-controlled Trial ("VITDAL@ICU")
Brief Title: VITdAL@ICU - Correction of Vitamin D Deficiency in Critically Ill Patients
Acronym: VITdAL@ICU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harald Dobnig, MD (Other)
Responsible Party: Sponsor-Investigator, Harald Dobnig, MD, Professor, Medical University of Graz
Organization: Medical University of Graz (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VITdAL@ICU - 19022010
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Critical Illness; Vitamin D Deficiency
MeSH Terms: conditions — Critical Illness; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol (Experimental)
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — loading dose of 540,000 IU of cholecalciferol via feeding tube or orally, then 5 monthly doses of 90,000 IU
  Arms: Cholecalciferol
Drug: Placebo — Matching placebo
  Other Names: herbal oil
  Arms: Placebo

SUMMARY:
Study hypothesis:

High-dose vitamin D leads to a shorter hospital stay in critically ill patients

Vitamin D deficient patients will be randomized to receive either 540,000 IU cholecalciferol or placebo.

DETAILED DESCRIPTION:
Inclusion criteria

* Age ≥18 years
* expected ICU stay ≥48 hours
* vitamin D deficiency: 25(OH)D ≤ 20 ng/ml
* feasibility of study drug application via nasogastric tube in cases where oral food intake is not possible

Exclusion criteria

* moribund patient expected to die within 24 hours
* hypercalcaemia (total calcium >2.65 OR ion. calcium >1.35 mmol/l)
* severely impaired gastrointestinal motility (ileus, residual gastric volume > 400 ml)
* known history of recent kidney stones (≤ 1 year)
* known granulomatous diseases (tuberculosis, sarcoidosis)
* pregnancy

Primary endpoint

* hospital stay (hours; starting from ICU admission) Secondary endpoints
* percentage of patients with 25(OH)D ≥ 30 ng/ml at day 7
* serum calcium; phosphorus; 25(OH)D; 1,25(OH)D; PTH; osteocalcin; bALP; TRAP; urinary calcium

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* expected ICU stay ≥48 hours
* vitamin D deficiency: 25(OH)D ≤ 20 ng/ml
* feasibility of study drug application via nasogastric tube in cases where oral food intake is not possible

Exclusion Criteria:

* moribund patient expected to die within 24 hours
* hypercalcaemia (total calcium >2.65 OR ion. calcium >1.35 mmol/l)
* severely impaired gastrointestinal motility (ileus, residual gastric volume > 400 ml)
* known history of recent kidney stones (≤ 1 year)
* known granulomatous diseases (tuberculosis, sarcoidosis)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2010-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | maximum 6 months
  The length of hospital stay will be compared between the two groups (starting from application of the study medication; end is defined as death of the patient or hospital discharge) Survivors and non-survivors will also be analysed separately. Stay in rehabilitation facilities will not be counted.

SECONDARY OUTCOMES:
25(OH)D levels | maximum 6 months
  serum 25(OH)D levels will be measured on day 0, 3 and 7
calcium levels | maximum 6 months
  serum calcium levels will be measured on day 0, 3 and 7
length of ICU stay starting from application of study medication | until patient's death or referral to another ward
duration of mechanical ventilation | starting from application of study medication
  duration of mechanical ventilation including CPAP/mask ventilation
hospital mortality, 28-day mortality, 6 month-mortality | maximum 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Dobnig, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Graz, Austria

REFERENCES:
- [Background] Lee P, Eisman JA, Center JR. Vitamin D deficiency in critically ill patients. N Engl J Med. 2009 Apr 30;360(18):1912-4. doi: 10.1056/NEJMc0809996. No abstract available. PMID 19403914
- [Background] Lucidarme O, Messai E, Mazzoni T, Arcade M, du Cheyron D. Incidence and risk factors of vitamin D deficiency in critically ill patients: results from a prospective observational study. Intensive Care Med. 2010 Sep;36(9):1609-11. doi: 10.1007/s00134-010-1875-8. Epub 2010 Apr 7. No abstract available. PMID 20373095
- [Background] Lee P, Nair P, Eisman JA, Center JR. Vitamin D deficiency in the intensive care unit: an invisible accomplice to morbidity and mortality? Intensive Care Med. 2009 Dec;35(12):2028-32. doi: 10.1007/s00134-009-1642-x. Epub 2009 Sep 15. PMID 19756497
- [Background] Mata-Granados JM, Vargas-Vasserot J, Ferreiro-Vera C, Luque de Castro MD, Pavon RG, Quesada Gomez JM. Evaluation of vitamin D endocrine system (VDES) status and response to treatment of patients in intensive care units (ICUs) using an on-line SPE-LC-MS/MS method. J Steroid Biochem Mol Biol. 2010 Jul;121(1-2):452-5. doi: 10.1016/j.jsbmb.2010.03.078. Epub 2010 Apr 21. PMID 20399267
- [Background] Krishnan A, Ochola J, Mundy J, Jones M, Kruger P, Duncan E, Venkatesh B. Acute fluid shifts influence the assessment of serum vitamin D status in critically ill patients. Crit Care. 2010;14(6):R216. doi: 10.1186/cc9341. Epub 2010 Nov 26. PMID 21110839
- [Background] Amrein K, Venkatesh B. Vitamin D and the critically ill patient. Curr Opin Clin Nutr Metab Care. 2012 Mar;15(2):188-93. doi: 10.1097/MCO.0b013e32834f0027. PMID 22186356
- [Background] Braun AB, Gibbons FK, Litonjua AA, Giovannucci E, Christopher KB. Low serum 25-hydroxyvitamin D at critical care initiation is associated with increased mortality. Crit Care Med. 2012 Jan;40(1):63-72. doi: 10.1097/CCM.0b013e31822d74f3. PMID 21926604
- [Background] Amrein K, Schnedl C, Berghold A, Pieber TR, Dobnig H. Correction of vitamin D deficiency in critically ill patients - VITdAL@ICU study protocol of a double-blind, placebo-controlled randomized clinical trial. BMC Endocr Disord. 2012 Nov 7;12:27. doi: 10.1186/1472-6823-12-27. PMID 23134762
- [Background] Amrein K, Zajic P, Schnedl C, Waltensdorfer A, Fruhwald S, Holl A, Purkart T, Wunsch G, Valentin T, Grisold A, Stojakovic T, Amrein S, Pieber TR, Dobnig H. Vitamin D status and its association with season, hospital and sepsis mortality in critical illness. Crit Care. 2014 Mar 24;18(2):R47. doi: 10.1186/cc13790. PMID 24661739
- [Derived] Schwetz V, Schnedl C, Urbanic-Purkart T, Trummer C, Dimai HP, Fahrleitner-Pammer A, Putz-Bankuti C, Christopher KB, Obermayer-Pietsch B, Pieber TR, Dobnig H, Amrein K. Effect of vitamin D3 on bone turnover markers in critical illness: post hoc analysis from the VITdAL-ICU study. Osteoporos Int. 2017 Dec;28(12):3347-3354. doi: 10.1007/s00198-017-4190-1. Epub 2017 Aug 25. PMID 28842727
- [Derived] Amrein K, Schnedl C, Holl A, Riedl R, Christopher KB, Pachler C, Urbanic Purkart T, Waltensdorfer A, Munch A, Warnkross H, Stojakovic T, Bisping E, Toller W, Smolle KH, Berghold A, Pieber TR, Dobnig H. Effect of high-dose vitamin D3 on hospital length of stay in critically ill patients with vitamin D deficiency: the VITdAL-ICU randomized clinical trial. JAMA. 2014 Oct 15;312(15):1520-30. doi: 10.1001/jama.2014.13204. PMID 25268295